CLINICAL TRIAL: NCT01633411
Title: Evaluation of Effect of CryoBalloon Focal Ablation System on Human Esophageal Barrett's Epithelium
Status: Completed | Type: Observational
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-0003.A
Record Dates: First submitted 2012-06-28; First posted 2012-07-04 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2015-04

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cohort A: Subjects in Cohort A will receive 6 seconds of treatment to dysplastic esophageal tissue using the Focal CryoBalloon Ablation System.
  Interventions: Device: Focal Cryoballoon Ablation System - 6 seconds
- Cohort B: Subjects in Cohort B will receive 8 seconds of treatment to dysplastic esophageal tissue using the Focal CryoBalloon Ablation System.
  Interventions: Device: Focal Cryoballoon Ablation System - 8 seconds
- Cohort C: Subjects in Cohort C will receive 10 seconds of treatment to dysplastic esophageal tissue using the Focal CryoBalloon Ablation System.
  Interventions: Device: CryoBalloon Focal Ablation System - 10 seconds

INTERVENTIONS:
Device: Focal Cryoballoon Ablation System - 6 seconds — Ablation of Barrett's Esophagus using a Focal Cryoballoon ablation catheter. The System is a Class II device "intended to be used as a cryosurgical tool for the destruction of unwanted tissue in the field of general surgery, specifically for endoscopic applications."
  Groups: Cohort A
Device: Focal Cryoballoon Ablation System - 8 seconds — Ablation of Barrett's Esophagus using a Focal Cryoballoon ablation catheter. The System is a Class II device "intended to be used as a cryosurgical tool for the destruction of unwanted tissue in the field of general surgery, specifically for endoscopic applications."
  Groups: Cohort B
Device: CryoBalloon Focal Ablation System - 10 seconds — Ablation of Barrett's Esophagus using the Focal CryoBalloon Ablation System. The System is a Class II device "intended to be used as a cryosurgical tool for the destruction of unwanted tissue in the field of general surgery, specifically for endoscopic applications".
  Groups: Cohort C

SUMMARY:
This is a feasibility study without a primary study hypothesis or statistical comparison.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, feasibility, and performance of the C2 Focal Cryoablation Device in patients with Barrett's Esophagus (BE). At 6 to 8 weeks, the patient will receive a follow-endoscopy to assess stricture formation along with biopsy samples taken.

Post-operative pain will be noted. Additionally, biopsy samples will be evaluated for the presence of residual Barrett's Esophagus. Through evaluation of the histological results, treatment parameters for the ablation of human esophageal epithelium will be better understood.

Evaluations include, but are not limited to the following:

* Deployment ease/scope compatibility.
* Device malfunctions.
* Time of catheter deployment.
* Adverse events.
* Stricture formation at 6 to 8 weeks.
* Patient Pain.
* Histological evaluation of treatment zone at 6 to 8 weeks for presence of residual Barrett's Esophagus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for ablation, EMR, and/or surveillance for BE (with or without dysplasia). Patient is 18 to 80 years of age at the time of consent (inclusive).
2. Patient has provided written Informed Consent (IC) using an Informed Consent Form (ICF) that has been approved by the Institution's reviewing IRB/EC.
3. Patient is willing and able to comply with all Clinical Investigation Plan (CIP) requirements.
4. Patient is deemed operable per standard institutional criteria.

Exclusion Criteria:

1. Patient with endoscopically active inflammation in the treatment zone
2. Esophageal stenosis preventing advancement of a therapeutic endoscope and/or within 4 cm of treatment zone.
3. Patient has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post treatment instructions or follow-up guidelines.
4. Patient refuses or is unable to provide written informed consent.
5. Patients that are pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Barrett's esophagus with or without dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Esophageal Stricture | 6 to 8 Weeks
  Stricture formation is defined as none, mild (non-circumferential stenosis allowing easy passage of diagnostic endoscope), moderate (circular stenosis allowing passage of diagnostic endoscope), and severe (any stenosis preventing the passage of a diagnostic scope).

SECONDARY OUTCOMES:
Post-procedure pain relative | Pre-ablation,12 hrs post ablation, 2 days (+ or - 1 day)
  A secondary objective of the study is to determine patient comfort post-procedure. Pain scores are measured on a numerical pain intensity scale (0 to 10). Patients is asked to score pain level in the treatment area and swallowing.
Presence of Residual Barrett's Esophagus | 6 to 8 weeks
  Esophageal tissue subjected to ablation via the CryoBalloon Focal Ablation System will be submitted for histological evaluation. The evaluation will include:
  1. detailed description of the presence of Barrett's Esophagus and/or squamous mucosa.
  2. estimate of percentage of residual Barrett's in each sample
  3. the detailed description of any residual injury at all levels within the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Bas L Weusten, MD, pHD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (8):
- United States (5):
  - University of Southern California, Los Angeles, California
  - John Hopkins, Baltimore, Maryland
  - Columbia Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
- Netherlands (3):
  - Academic Medical Center Amsterdam, Amsterdam
  - St. Antonius Hospital, Nieuwegein
  - Universitair Medisch Centrum Utrecht, Utrecht

REFERENCES:
- [Background] Friedland S, Triadafilopoulos G. A novel device for ablation of abnormal esophageal mucosa (with video). Gastrointest Endosc. 2011 Jul;74(1):182-8. doi: 10.1016/j.gie.2011.03.1119. Epub 2011 Apr 30. PMID 21531411
- See also: Related Info — http://pentaxmedical.com